CLINICAL TRIAL: NCT02041845
Title: A Randomized Phase II Study Comparing Two Schedules of Hyperfractionated Thoracic Radiotherapy in Limited Disease Small Cell Lung Cancer
Brief Title: Two Schedules of Hyperfractionated Thoracic Radiotherapy in Limited Disease Small Cell Lung Cancer
Acronym: THORA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/2163
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Radiotherapy; Radiotherapy dosage; Dose fractionation; Radiotherapy, image-guided; Thorax
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 3D conformal thoracic radiotherapy at a total dose of 45 Gy in 30 fractions, 2 fractions per day, 5 days a week
  Interventions: Radiation: 45 Gy in 30 fractions
- B (Experimental): 3D conformal thoracic radiotherapy at a total dose of 60 Gy in 40 fractions, 2 fractions per day, 5 days a week
  Interventions: Radiation: 60 Gy in 40 fractions

INTERVENTIONS:
Radiation: 45 Gy in 30 fractions — 3D conformal thoracic radiotherapy at a total dose of 45 Gy in 30 fractions, 2 fractions per day, 5 days a week
  Arms: A
Radiation: 60 Gy in 40 fractions — 3D conformal thoracic radiotherapy at a total dose of 60 Gy in 40 fractions, 2 fractions per day, 5 days a week. If doses to organs at risk exceed normal tissue tolerance, the dose may be lowered to a minimum of 54 Gy.
  Arms: B

SUMMARY:
The majority of patients with limited disease small cell lung cancer (SCLC) experience recurrent disease despite receiving concurrent chemoradiotherapy. New agents and dose-escalation of chemotherapy have not provided a survival benefit. Local failure accounts for high proportion of recurrences. Improved thoracic radiotherapy (TRT) might increase local control and thus reduce the recurrence rate and prolong survival. Positron emission tomography (PET CT) is better for staging of SCLC than computer tomography (CT) and bone scan. More precise localization of tumors leads to more accurate definition of target volumes for TRT and reduce the radiation dose to normal tissue. A large proportion of patients relapse and die within one and two year after therapy. Few patients survive longer than three years. Thus, two-year survival is considered a clinically highly relevant measure of efficacy.

The aim of this study is to compare two schedules of TRT with respect to local control, progression free survival, overall survival, toxicity and health-related quality of life. In addition patients who have the best outcomes and tolerate chemoradiotherapy will be characterized (e.g. clinical characteristics, blood biomarkers, body composition).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small-cell lung cancer (SCLC)
* Limited disease (stage II-III)
* Stage I if ineligible for surgery
* Eastern Cooperative Oncology Group (ECOG) Performance 0-2
* Measureable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Adequate organ function defined as: (a) Serum serum alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN); (b) Total serum bilirubin ≤ 1.5 x ULN; (c) Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; (d) Platelets ≥ 100 x 109/L; (e) Creatinine < 100 µmol/L and calculated creatinine-clearance > 50 ml/min. If calculated creatinine-clearance is < 50 ml/min, an ethylene diamine tetra-acetic acid (EDTA) clearance should be performed.
* Pulmonary function: Forced Expiratory Volume in One Second (FEV1) > 1 l or 30 % of predicted value and diffusing capacity of the lungs for carbon monoxide (DLCO) > 30 % of predicted value
* All fertile patients should use safe contraception
* Written informed consent

Exclusion Criteria:

* prior systemic therapy for small-cell lung cancer
* Previous radiotherapy to the thorax
* malignant cells in pericardial or pleural fluid (at least one sample should be analysed if pleural fluid is present
* serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study treatment
* conditions - medical, social, psychological - which could prevent adequate information and follow-up
* clinically active cancer other than SCLC. Hormonal therapy for prostate cancer or breast cancer and basocellular carcinoma of the skin is allowed
* pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
survival | 2 years
  measured for all patients from the date of the first day of the first course of chemotherapy until the date of death from any cause (or last contact/observation if lost to follow-up - or the follow-up is completed before all patients die).

SECONDARY OUTCOMES:
progression free survival (PFS) | 2 years
  measured for all patients from the date of the first day of the first course of PE to the first date of objective progression (according to RECIST 1.1) of disease or of death from any cause. For each patient who has not died or has non-progression at the cut-off date for the analysis, PFS will be censored at the date of the patient's last tumor assessment prior to the cut-off date. Statistical survival analyses will be done with Kaplan Meier. Log rank test will be used for comparing groups.
Local control | 2 years
  Proportion of all patients who experience disease recurrence within radiotherapy fields assessed by comparing dose plans and follow-up CT scans.
overall survival | 3 years
  measured for all patients from the date of the first day of the first course of chemotherapy until the date of death from any cause (or last contact/observation if lost to follow-up - or the follow-up is completed before all patients die).
toxicity | 2 years
  assessed for all patients receiving at least one course of chemotherapy from reported blood values and adverse event. Classified and graded according to CTCAE 4.0. Compared using Pearson's Chi-square and Fischer's exact tests.
health related quality of life (HRQoL) | From baseline, before and after radiotherapy and then at follow-up every 3 months until 24 months after start of chemotherapy. Then every 6 months until 5 year after start of therapy
  assessed from completed questionnaires. Patients will report HRQoL on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 and the lung cancer specific module LC13. The QLQ-C30 measures fundamental aspects of HRQoL and symptoms commonly reported by cancer patients in general, the LC13 measures symptoms commonly associated with lung cancer and its treatment.
  All HRQoL scores will be transformed to a scale from 0 to 100 according to the EORTC scoring manual. A difference in mean scores of >10 is considered clinically relevant. For group comparisons of baseline scores during and after chemotherapy, and changes in scores from baseline, the Mann-Whitney test will be used. Primary HRQoL-endpoints are dysphagia and dyspnea.

OTHER OUTCOMES:
Exploratory analyses of associations between characteristics and blood biomarkers - and outcomes of therapy | 3 years
  All patients will be included in these analyses. Blood will be collected, the study group will define which markers to analyze when all patients have been enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn H Grønberg, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (22):
- Denmark (2):
  - Rigshospitalet København, Copenhagen
  - Odense University Hospital, Odense
- Norway (14):
  - Ålesund sykehus, Ålesund
  - Haukeland Universitetssykehus, Bergen
  - Vestre Viken HF, Drammen Sykehus, Drammen
  - Førde Sentralsykehus, Førde
  - Sykehuset Innlandet Gjøvik, Gjøvik
  - Haugesund sykehus, Haugesund
  - Sykehuset Levanger, Levanger
  - Sykehuset Namsos, Namsos
  - Akershus Universitetssykehus, Oslo
  - Oslo Universitetssykehus, Radiumhospitalet, Oslo
  - Sykehuset Østfold (Kalnes/Sarpsborg), Sarpsborg
  - Universitetssjukehuset i Stavanger, Stavanger
  - University Hospital of North Norway, Pulmonology Department, Tromsø
  - Cancer Clinic at St. Olavs Hospital, Trondheim
- Sweden (6):
  - Gävle Sjukhus, Gävle
  - Sahlgrenska Sjukehuset, Gothenburg
  - Skånes universitetssjukhus, Lund
  - Universitetssjukehuset i Ôrebro, Örebro
  - Karolinska University Hospital, Stockholm
  - Norrlands Universitetssjukehus, Umeå

REFERENCES:
- [Result] Gronberg BH, Killingberg KT, Flotten O, Brustugun OT, Hornslien K, Madebo T, Langer SW, Schytte T, Nyman J, Risum S, Tsakonas G, Engleson J, Halvorsen TO. High-dose versus standard-dose twice-daily thoracic radiotherapy for patients with limited stage small-cell lung cancer: an open-label, randomised, phase 2 trial. Lancet Oncol. 2021 Mar;22(3):321-331. doi: 10.1016/S1470-2045(20)30742-7. PMID 33662285
- [Derived] Gronberg BH, Killingberg KT, Flotten O, Bjaanaes MM, Brustugun OT, Madebo T, Langer SW, Risumlund SL, Schytte T, Helbekkmo N, Neumann K, Yksnoy O, Engleson J, Fluge S, Naustdal T, Giske LE, Nyman J, Tsakonas G, Halvorsen TO. High-Dose Versus Standard-Dose Twice-Daily Thoracic Radiotherapy in Limited-Stage SCLC: Final Survival Data, Long-Term Toxicity, and Relapse Patterns in a Randomized, Open-Label, Phase II Trial. J Thorac Oncol. 2025 Aug;20(8):1108-1119. doi: 10.1016/j.jtho.2025.04.007. Epub 2025 Apr 19. PMID 40258573
- [Derived] Taranova E, Aanerud M, Halvorsen TO, Killingberg KT, Slaaen M, Gronberg BH. Associations Between Patient-Reported Nutritional Status, Toxicity, and Survival in Limited-Stage SCLC. JTO Clin Res Rep. 2024 Nov 12;6(1):100764. doi: 10.1016/j.jtocrr.2024.100764. eCollection 2025 Jan. PMID 39802818
- [Derived] Killingberg KT, Gronberg BH, Slaaen M, Kirkevold O, Halvorsen TO. Treatment Outcomes of Older Participants in a Randomized Trial Comparing Two Schedules of Twice-Daily Thoracic Radiotherapy in Limited-Stage SCLC. J Thorac Oncol. 2023 Jun;18(6):803-812. doi: 10.1016/j.jtho.2023.01.012. Epub 2023 Jan 27. PMID 36716960
- [Derived] Killingberg KT, Halvorsen TO, Flotten O, Brustugun OT, Langer SW, Nyman J, Hornslien K, Madebo T, Schytte T, Risum S, Tsakonas G, Engleson J, Gronberg BH. Patient-reported health-related quality of life from a randomized phase II trial comparing standard-dose with high-dose twice daily thoracic radiotherapy in limited stage small-cell lung cancer. Lung Cancer. 2022 Apr;166:49-57. doi: 10.1016/j.lungcan.2022.02.002. Epub 2022 Feb 8. PMID 35183991